CLINICAL TRIAL: NCT05199220
Title: Epidemiology of Injuries During Crossfit Practice : a Prospective Cohort Study at Reunion Island
Brief Title: Epidemiology of Injuries During Crossfit Practice
Acronym: EPITRAUMA-CF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/26
Record Dates: First submitted 2021-12-06; First posted 2022-01-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2021-11

CONDITIONS: Sport Injury
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Participant must complete a questionnaire about injury during crossfit practice
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participant must complete a questionnaire about injury during crossfit practice

SUMMARY:
This study aims to precisely describe epidemiology of injuries than occur during practice of crossfit. Each participant will complete questionnaires in order to identify injuries. The first questionnaire will be completed at the moment of the inclusion and the second questionnaire will be completed if participant has injuries every 3 months until month 12.

ELIGIBILITY:
Inclusion Criteria:

* person affiliated to a crossfit structure at Reunion Island at the beginning of the study
* personne who agrees to participate in the study

Exclusion Criteria:

* person under tutorship or curatorship,
* person whose the initial questionnaire initial is complete,
* person who can neither read nor write french.
* person planning to leave Reunion Island within 12 months after enrolment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult who practices crosffit must be included in Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Location of injury by questionnaire | at month 3
  the location of the injury on the body must be specified
laterality of injury by questionnaire | at month 3
  Laterality of injury must be precised if to be at right or left
mechanism of injury by questionnaire | at month 3
  it will be identified as a traumatic injury or an overuse. Traumatic injury is due to an acute identified event. An overuse is due to repetitive train injury.
circumstance of injury occurence by questionnaire | at month 3
  circumstance is defined as when occurs injury : suddenly or gradually
injury relapse or not | at month 3
  injury relapse is classified as early relapse if occurs within 2 months after the healing, as late relapse if occurs from 2 months to 12 months after the healing or as very late relapse if occurs after more 12 months.
diagnosis of injury | at month 3
  diagnosis will be classified according to the OSICS 10 classification
record of exposure to injury | at month 3
  Training volume will be recorded by level of practice (leisure practice, club practice and competition practice)

CONTACTS AND LOCATIONS:
Locations (1):
- Crosffit Structure, Saint-Pierre, Reunion